CLINICAL TRIAL: NCT01383447
Title: A Phase 1/2 Study of SNDX-275 in Combination With Imatinib for Relapsed/Refractory Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
Brief Title: Entinostat And Imatinib Mesylate In Treating Patients With Relapsed or Refractory Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was halted prematurely by the NCI for low accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2010-02202; J1023; U01CA070095 (NIH)
Record Dates: First submitted 2011-05-05; First posted 2011-06-28 (Estimated); Results first posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-07

CONDITIONS: Philadelphia Chromosome Positive Adult Precursor Acute Lymphoblastic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — entinostat; Imatinib Mesylate; Blotting, Western; Immunohistochemistry; Flow Cytometry; Polymerase Chain Reaction; Chromatography, High Pressure Liquid; Mass Spectrometry

ARMS (1):
- Treatment (entinostat and imatinib mesylate) (Experimental): Patients receive entinostat PO daily on days 1, 8, 15, and 22 and imatinib mesylate PO twice daily on days 1-28 (days 4-28 of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: entinostat; Drug: imatinib mesylate; Other: laboratory biomarker analysis; Other: pharmacological study; Genetic: western blotting; Other: immunohistochemistry staining method; Other: flow cytometry; Genetic: polymerase chain reaction; Other: high performance liquid chromatography; Other: mass spectrometry

INTERVENTIONS:
Drug: entinostat — Given PO
  Other Names: HDAC inhibitor SNDX-275; SNDX-275
Drug: imatinib mesylate — Given PO
  Other Names: CGP 57148; Gleevec; Glivec
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Genetic: western blotting — Correlative studies
  Other Names: Blotting, Western; Western Blot
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Other: flow cytometry — Correlative studies
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR
Other: high performance liquid chromatography — Correlative studies
  Other Names: HPLC
Other: mass spectrometry — Correlative studies

SUMMARY:
This phase I/II trial is studying the side effects and best dose of entinostat when given together with imatinib mesylate and to see how well it works in treating patients with relapsed or refractory Philadelphia chromosome-positive acute lymphoblastic leukemia. Entinostat and imatinib mesylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of entinostat when given in combination with imatinib (matinib mesylate).

SECONDARY OBJECTIVES:

I. To estimate the rate of complete response (CR) for patients greater ≥ 18 years of age with relapsed/refractory Ph+ ALL treated with a combination of entinostat and imatinib.

II. To estimate the 1 year progression free survival (PFS) for patients greater ≥ 18 years of age with relapsed/refractory Ph+ ALL treated with a combination of entinostat and imatinib III. To describe the comparative pharmacokinetics (PK) and pharmacodynamics (PD) of entinostat when administered alone vs. in combination with imatinib.

IV. To assess the predictive value of levels of flow cytometric minimal residual disease (MRD) on duration of progression free survival for the study population.

OUTLINE: This is a phase I, dose-escalation study of entinostat followed by a phase II study.

Patients receive entinostat orally (PO) daily on days 1, 8, 15, and 22 and imatinib mesylate PO twice daily on days 1-28 (days 4-28 of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed BCR-ABL1 associated (Ph+) acute lymphoblastic leukemia (ALL) with primary refractory or relapsed disease; demonstration of BCR-ABL1 in leukemia cells by one or more of the following is required: t(9;22)(q34;q11.2) cytogenetics; FISH for BCR-ABL1 fusion; RT-PCR for BCR-ABL1 fusion
* Prior treatment with tyrosine kinase inhibitors (including imatinib, nilotinib and/or dasatinib) is allowed, although patients must be off any tyrosine kinase inhibitor for a minimum of 72 hours prior to beginning protocol therapy
* ECOG performance status of 0, 1 or 2
* Total WBC =< 150,000 with no evidence for ongoing or impending leukostasis
* Total bilirubin =< 2.0 mg/dL unless elevated due to Gilbert's, hemolysis or leukemic infiltration
* Aspartate transaminase (AST)/alanine transaminase (ALT) =< 2.5 × upper limit of normal (ULN) unless due to leukemic infiltration
* Serum creatinine =< 2.0 mg/dL or creatinine clearance > 50 ml/min
* Left ventricular ejection fraction (LVEF) >= 45% as measured by echocardiogram (ECHO) or MUGA
* Patients who have undergone stem cell transplantation (SCT), autologous or allogeneic, are eligible provided that they are > 4 weeks from stem cell infusion, have no active GVHD, and meet other eligibility criteria
* Patients who fail primary induction therapy or relapse after achieving complete remission (CR) are eligible if they are > 3 weeks off cytotoxic chemotherapy and > 2 weeks off radiation therapy; patients must be off biologic therapies including hematopoietic growth factors > 1 week; if using hydroxyurea (HU), steroids, or other non-cytotoxics for blast count control, patient must be off for > 24 hrs before starting protocol therapy; patients must have recovered from all acute toxicities from any previous therapy
* Female patients of childbearing age must have negative pregnancy test; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Active CNS leukemia; patients with known previous CNS leukemia may continue to receive intrathecal therapy with ara-C, methotrexate, and/or thiotepa plus steroids as prophylaxis against reactivation of previous CNS disease
* Patients may not have received previous treatment with entinostat or other HDAC inhibitors
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to entinostat or other agents used in study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active untreated infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with entinostat
* HIV-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Brown, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Entinostat and Imatinib Mesylate)
Started | 2
Completed | 0
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Entinostat and Imatinib Mesylate)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Entinostat When Given in Combination With Imatinib Mesylate
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting.
Time Frame: Up to 30 days post-treatment
Population: This study was halted prematurely by the NCI for low accrual. No results were analyzed.
Arm/Group | Treatment (Entinostat and Imatinib Mesylate)
Number analyzed (Participants) | 0

2. Secondary Outcome: Rate of Complete Response (CR) for Adults With Relapsed/Refractory Ph+ ALL Treated With a Combination of Entinostat (at the Dose Determined in Phase 1) and Imatinib Mesylate
Time Frame: Up to 30 days post-treatment
Population: This study was halted prematurely by the NCI for low accrual. No results were analyzed.
Arm/Group | Treatment (Entinostat and Imatinib Mesylate)
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression Free Survival (PFS) for Adults With Relapsed/Refractory Ph+ ALL Treated With Combination of Entinostat and Imatinib Mesylate
Description: The Kaplan-Meier estimator will be used to estimate PFS with a 95% confidence interval from study entry.
Time Frame: At 1 year
Population: This study was halted prematurely by the NCI for low accrual. No results were analyzed.
Arm/Group | Treatment (Entinostat and Imatinib Mesylate)
Number analyzed (Participants) | 0

4. Secondary Outcome: Comparative Pharmacokinetics (PK) and Pharmacodynamics (PD) of Entinostat Alone vs. Entinostat Plus Imatinib Mesylate
Description: Entinostat concentrations will be compared when administered alone or in combination with imatinib by paired Student's t test (day 4 vs 11 concentrations) or Wilcoxon signed rank tests as appropriate. Association between exposure parameters and PD endpoints (e.g., apoptosis, histone acetylation, BCR-ABL expression) will be assessed using Fisher's exact tests or Wilcoxon rank sum tests as appropriate.
Time Frame: Day 4 and 11
Population: This study was halted prematurely by the NCI for low accrual. No results were analyzed.
Arm/Group | Treatment (Entinostat and Imatinib Mesylate)
Number analyzed (Participants) | 0

5. Secondary Outcome: Predictive Values of Levels of Flow Cytometric Minimal Residual Disease (MRD) on Duration of Progression Free Survival for the Study Population
Description: Kaplan-Meier PFS curves and cumulative incidence of progression curves will be generated for patients above vs. below each threshold, and log rank will be used to compare the curves.
Time Frame: Day 29
Population: This study was halted prematurely by the NCI for low accrual. No results were analyzed.
Arm/Group | Treatment (Entinostat and Imatinib Mesylate)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Entinostat and Imatinib Mesylate)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Entinostat and Imatinib Mesylate) (N=2)
Edema: lower limb (General disorders) | 1
nausea (Gastrointestinal disorders) | 1
Insomnia (Psychiatric disorders) | 1
Pain: bone marrow site (Musculoskeletal and connective tissue disorders) | 1
Fatigue (General disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less